CLINICAL TRIAL: NCT02778464
Title: PREGCAL: Pilot Study to Assess Faecal Calprotectin as a Potential Non-invasive Inflammatory Marker in Pregnancy and Inflammatory Bowel Disease
Brief Title: Faecal Calprotectin as a Potential Non-invasive Inflammatory Marker in Pregnancy and Inflammatory Bowel Disease
Acronym: PREGCAL
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015GAS78
Record Dates: First submitted 2016-04-05; First posted 2016-05-19 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Inflammatory Bowel Disease (IBD); Crohn's Disease (CD); Ulcerative Colitis (UC); Pregnancy
Keywords: Inflammatory Bowel Disease; Pregnancy; Stool markers; Calprotectin; Faecal S100A12 (f-SA12); Faecal calprotectin (f-Cp)
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Faecal calprotectin, faecal S100A12, serum S100 and serum calprotectin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group A: Female IBD and RA (non-pregnant): This group will be asked to provide three blood samples, one in each trimester. Stool samples are expected to average 8-10 per participant. All diaries and stool sample consumables for disease activity will be issued at the initial visit. Bloods will be obtained at a hospital visit. Stool samples due between hospital visits will be obtained according to protocol to minimise pre-analytical variance.
- Group B: Female IBD: This group will be asked to provide three blood samples, one in each trimester. Stool samples are expected to average 8-10 per participant. All diaries and stool sample consumables for disease activity will be issued at the initial visit. Bloods will be obtained at a hospital visit. Stool samples due between hospital visits will be obtained according to protocol to minimise pre-analytical variance.
- Group C: Female - Healthy Pregnant: This group will be asked to provide three blood samples, one in each trimester. Stool samples are expected to average 8-10 per participant. All stool sample consumables will be issued at the initial visit. Bloods will be obtained at a hospital visit. Stool samples due between hospital visits will be obtained according to protocol to minimise pre-analytical variance.
- Group D: Female - RA Pregnant: This group will be asked to provide three blood samples, one in each trimester. Stool samples are expected to average 8-10 per participant. All stool sample consumables will be issued at the initial visit. Bloods will be obtained at a hospital visit. Stool samples due between hospital visits will be obtained according to protocol to minimise pre-analytical variance.

SUMMARY:
When women with rheumatoid arthritis become pregnant 75% of them will go into remission, despite stopping medication. This phenomenon is not well understood and is not seen in other inflammatory conditions. Once they give birth they often relapse. Bacteria in the stool and inside the gut have the ability to effect the immune system and some beneficial bacteria are known to down regulate inflammatory components of the immune system. Gut bacteria are also known to alter significantly during pregnancy and in other inflammatory conditions there are low levels of beneficial bacteria associated with diseases like ulcerative colitis. There is significant crossover between rheumatoid arthritis and inflammatory bowel disease with similar arthritic symptoms and mechanisms of inflammation. There is very limited investigation of gut bacteria and rheumatoid arthritis, but some animal work has shown that treatment with probiotics and prebiotics can improve the condition. The aim of this study is to examine the bacteria in the stool of women who are pregnant with rheumatoid arthritis and identify any significant bacteria changes that might be used to direct future research.

DETAILED DESCRIPTION:
Pregnancy has an interesting and different impact on inflammatory conditions that have much in common immunologically. In inflammatory bowel disease 33% will deteriorate, 33% will remain stable and 33% will improve. In rheumatoid arthritis 75% of women will improve. Gut microbiota alters significantly in pregnancy as do predominant immunological pathways and relapse post-partum is swift. Research on intestinal microbiota in women with inflammatory conditions is scant. The high remission rate in pregnancy gives us a unique opportunity to study the microbiota for changing patterns that could be identified in the future as potential therapeutic targets.

The study aims to identify any bacterial changes from pre-conception through pregnancy to post-partum and comparing women who relapse with rheumatoid arthritis to those who remain in remission.

Clinical condition will be assessed and stool and serum samples will be obtained from women during each trimester during pregnancy for analysis of serum and fecal biomarkers and for microbiota 16S rRNA (ribosomal ribonucleic acid) techniques. Group-specific 16S rRNA-targeted oligonucleotide probes labeled with the fluorescent dye Cy3 will be used for enumerating bacteria. The probes used will determine bifidobacteria, bacteroides, clostridia (Clostridium perfringens/histolyticum sub. Grp.), eubacterium recale-C histolyticum sub gp., agrobacterium rimae - Collinsella-Eggerthella lenta sub. Gp., Lactobacillus/Enterococcus spp., desulfovibrio spp., Faecalibacterium prausnitzii and Escherichia coli, interferon-gamma and Interleukin 10 (IL-10). Total bacteria will be enumerated using flow cytometry techniques.

The outcomes of this project would help identify microbiota patterns and bacteria species that are beneficial in rheumatoid arthritis and could be targets for potential gut immunomodulation therapy in the future to prolong periods of remissions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women (i.e. no-IBD and no significant comorbidities). pregnant IBD and rheumatoid women with any class of disease activity, non-pregnant IBD women and Rheumatoid arthritis women aged between 18 and 40.

Exclusion Criteria:

* Coeliac disease
* Familial adenomatous polyposis and hereditary nonpolyposis
* Rheumatoid arthritis (in healthy group or IBD groups)
* Irritable bowel syndrome (ROME III criteria)
* Lactose intolerance
* Other connective tissue inflammatory diseases
* Active infection
* NSAID, aspirin or anticoagulant us,
* Recipients of antibiotics in under 4 weeks of initial trial participation
* Women on the oral contraceptive pill

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women are the basis of this study, both with and without IBD to be able to meet the primary objective. As a feasibility study, there is no data on what levels are to be expected in pregnant women and if those results may vary at different stage of pregnancy. The investigators have chosen a small population size that reflects their anticipated recruitment levels of pregnant IBD patients over 2 years in the West Midlands. The investigators would expect to see 2-3 pregnant IBD patients per annum. Across 7 identified collaborating sites to take part the investigators anticipate there to be between 30-42 patients eligible over a 2 year period.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Measure faecal calprotectin in pregnant IBD patients and compare to healthy controls | 24 Months
  Measuring faecal calprotectin in pregnant IBD patients and comparing to healthy controls in a feasibility study will see if it may be of use as a marker of intestinal inflammation during pregnancy.

SECONDARY OUTCOMES:
Assess elevated f-CP in pregnant, healthy patients | 24 months
  If pregnant healthy patients have elevated f-CP levels outwith the standard range for normal. If they do not, then demonstrating that against an IBD cohort may mean that they can be used as surrogate markers of inflammation even in pregnancy
Assess elevated f-CP levels in IBD patients | 24 months
  If the f-CP levels are raised if they compare with those of IBD patients, and therefore the marker becomes unreliable or if there is a difference, could lead to a larger national study to quantify sensitivity and specificity of the test in this group of patients
Measure serum calprotectin levels in faeces | 24 Months
  Measurements for serum calprotectin will also be taken to compare to faecal levels and see if they correlate to fluctuate at different times during pregnancy
Assess elevated f-SA12 levels in pregnant, healthy patients | 24 months
  If pregnant healthy patients have elevated f-SA12 levels outwith the standard range for normal. If they do not, then demonstrating that against an IBD cohort may mean that they can be used as surrogate markers of inflammation even in pregnancy
Assess elevated f-SA12 levels in IBD patients | 24 Months
  If the f-SA12 levels are raised if they compare with those of IBD patients, and therefore the marker becomes unreliable or if there is a difference, could lead to a larger national study to quantify sensitivity and specificity of the test in this group of patients

CONTACTS AND LOCATIONS:
Overall Officials: Helen Steed, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No